CLINICAL TRIAL: NCT05984173
Title: the Role of Vitamin E in Reducing Incidence of Dry Socket in Female Patients. A Randomized Clinical Trial
Brief Title: Role of Vitamin E in Reducing Dry Socket
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7132023asu
Record Dates: First submitted 2023-07-22; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-01

CONDITIONS: Dry Socket
Keywords: dry socket
MeSH Terms: conditions — Dry Socket | interventions — Tocopherols

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial two groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patients received vitamin E inside the socket after extraction (study group)
  Interventions: Drug: Vitamin E application
- control (No Intervention): patients didn't receive vitamin E after extraction (control group).

INTERVENTIONS:
Drug: Vitamin E application — patients received vitamin E inside the socket after extraction
  Other Names: tocopherol
  Arms: study group

SUMMARY:
90 female patients seeking extraction of a single tooth in the lower posterior region were divided randomly into 45 patients received vitamin E inside the socket after extraction (study group) and 45 patients didn't receive vitamin E after extraction (control group).

DETAILED DESCRIPTION:
I. Patient Selection and Grouping:

This study was conducted on a total number of 90 female patients seeking extraction of a single tooth in the lower posterior region, selected from those attending the outpatient clinic of the oral and maxillofacial surgery department in the faculty of dentistry, Ain Shams University and Misr University for Science & Technology, Egypt as divided randomly into 45 patients received vitamin E inside the socket after extraction (study group) and 45 patients didn't receive vitamin E after extraction (control group).

II. Sample Size Calculation:

In the prior assessment of the article by Haraji et al. (Effects of Intra-alveolar Placement of 0.2% Chlorhexidine Bioadhesive Gel on Dry Socket Incidence and Postsurgical Pain: A Double-Blind Split-Mouth Randomized Controlled Clinical Trial) and setting alpha at 0.05 and Beta at 0.8 the data showed that the minimum number of patients to be included in each group was 18.

III. Blinding\Masking:

Blinding of biostatistician was achieved while blinding of participants and operator wasn't possible as the operator is the outcome assessor.

IV. Research Ethics Approval:

The research was reviewed by the Research Ethics Committee (REC) of the Faculty of Dentistry, Ain Shams University.

V. Preoperative Assessment:

1. Patient Evaluation:

   Each female has been evaluated for the following:

   A. Medical History:

   Full medical history was taken to exclude any patient according to the exclusion criteria.

   B. Dental History:

   Full dental history was taken including the history of previous incidences of dry socket.

   C. Chief Complaint All patients were asked about the current dental chief complaint to exclude any patient who needed dental treatment other than extraction.
2. Clinical Examination:

   A. Extra-Oral Examination:

   All patients were examined by the operator including facial appearance and facial bone.

   B. Intra-Oral Examination:

   This examination included:
   * General examination of oral health, checking the teeth adjacent to the extracted tooth and oral hard and soft tissues.
   * Examination of extracted tooth including tenderness and mobility tests.
3. Radiographic Assessment Radiographic assessment was done using a periapical radiograph to examine the surrounding bone, exclude any pathological lesion, and detect the location of the inferior alveolar canal, especially during extraction of lower third molars.
4. Photography:

   Intra-oral Photographs were taken before establishing the surgical procedure. Figure (1)
5. Surgical Preparation:

A. Anesthetic Protocol:

The extraction procedures were done under local anesthesia using 4% articaine solution with adrenaline 1:100,000, as 1.2 ml for Inferior Alveolar Nerve block (IANB), 0.3 ml for lingual nerve block and 0.3 ml for long buccal nerve block on the side of the extraction.

B. Preparation of Gel Foam and Vitamin E:

A piece of gel foam was cut into 1 X1 cm2.

C. Extraction Procedure:

* All extractions were performed by the same surgeon using standard English-Style Vertical Hinge forceps in a standardized buccolingual technique for socket expansion.
* The extraction procedures were done simply using forceps or elevators without raising mucoperiosteal flaps or anything that make the procedure surgical. Figure (2)

D. Packing of the Gel Foam:

The prepared gel foam was packed inside the socket to be covering the walls of the socket and not be oversized.

E. Suture with Figure 8:

A horizontal Figure 8 suture was applied for stabilization. Figure (3)

F. Post-Operative Instructions:

* Keep biting on the gauze for 1 hour.
* Avoid eating or drinking hot stuff on the first post-extraction day.
* Soft and cold food can be consumed after 2 hours on the other side.
* Avoid rinsing for the next 24 hours after extraction.
* Rinsing the mouth with warm saline 3 times daily on the 2nd day and continued for 5 days.
* Avoid smoking.
* Rest and avoid strenuous activities for the remainder of the day.
* Patients were given a prescription for Diclofenac Potassium to be used twice daily for three days.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 30-50 years of age.
* Patients with single tooth in the lower posterior region need simple extraction.
* Compliance with all requirements in the study and signing the informed consent.

Exclusion Criteria:

* Patients with any medical condition that may influence the outcome (uncontrolled diabetes, Hyperparathyroidism, Hyperthyroidism, Cushing's disease, Paget's disease, Glucocorticoids).
* Vulnerable groups (children, pregnant women, elderly people, malnourished people, prisoners, migrants, and refugees).
* Patients with systemic disease affecting bone healing (osteoporosis, Rickets, and osteomalacia).
* Chronic Patients on medications known to affect the periodontal status (calcium antagonists, anticonvulsive, immunosuppressive, anti-inflammatory medications).
* Patients with a history of bisphosphonate use.
* Pathologic lesions in the site of extraction.
* Lactating mothers.
* Smoking patients.
* Patients currently on radiotherapy and or chemotherapy treatment.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only biological female because estrogen is limiting factor
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Decrease of incidence of dry socket and pain | one week
  Evaluation of patient satisfaction and pain was done and recorded according to VAS which is a scale from 1-10. patient mention degree of pain on this scale

CONTACTS AND LOCATIONS:
Overall Officials: mohamed diaa, Study Director — Ain shams
Locations (1):
- Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Not planning to share

REFERENCES:
- [Result] Blum IR. Contemporary views on dry socket (alveolar osteitis): a clinical appraisal of standardization, aetiopathogenesis and management: a critical review. Int J Oral Maxillofac Surg. 2002 Jun;31(3):309-17. doi: 10.1054/ijom.2002.0263. PMID 12190139